CLINICAL TRIAL: NCT00546000
Title: A Multi-Center, Open-Label Study to Evaluate the Effect of ALTANA Inc's Cutivate (Fluticasone Propionate) Lotion 0.05% on the Hypothalmic Pituitary Adrenal (HPA) Axis in the Treatment of Atopic Dermatitis in a Pediatric Population
Brief Title: Cutivate Lotion HPA Axis Pediatric Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALT 0434-01-01
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Receive between 22 and 29 days of Cutivate lotion treatment
  Interventions: Drug: Fluticasone propionate 0.05% lotion

INTERVENTIONS:
Drug: Fluticasone propionate 0.05% lotion — Daily applications

SUMMARY:
A multi-center, open-label, Phase IV, unblinded study using Cutivate (fluticasone propionate, 0.05%)lotion and it's possible effects on the HPA axis of infants diagnosed with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are 3-12 months of age
* Subjects diagnosed with Atopic Dermatitis (AD) and have ≥35% of Body Surface Area
* Subjects meet protocol specific AD signs and symptom severity score

Exclusion Criteria:

* Subjects with conditions effecting the HPA Axis
* Subjects with clinically significant systemic disease
* Subjects who require treatment with systemic or topical retinoids during the study
* Subjects who have been treated with various chronic therapies identified in the protocol
* Subjects who have received other investigational drug treatment within 30 days prior to study entry

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Fleischer Jr., M.D., Principal Investigator — Wake Forest University Health Sciences; Lawrence F. Eichenfield, MD, Principal Investigator — Rady Children's Hospital, San Diego; Elizabeth Connelly, MD, Principal Investigator — University of Miami; Craig L. Leonardi, MD, Principal Investigator — Central Dermatology; Lawrence Parish, MD, Principal Investigator — Paddington Testing Company, Inc; Adelaide A Hebert, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Sharon Raimer, MD, Principal Investigator — University of Texas Medical Branch, Galveston; Kenneth E. Bloom, MD, Principal Investigator — Dermatology Center for Children and Young Adults; David L Kaplan, MD, Principal Investigator — Adult & Pediatric Dermatology; Stephen W. Shewmake, M.D., Principal Investigator — Centre for Health Care Medical Associates
Locations (10):
- United States (10):
  - Centre for Health Care Medical Associates, Poway, California
  - Rady Children's Hospital, San Diego, San Diego, California
  - University of Miami, Dept. of Dermatology, Miami, Florida
  - Adult & Pediatric Dermatology, Overland Park, Kansas
  - Dermatology Center for Children and Young Adults, Eagan, Minnesota
  - Central Dermatology, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Paddington Testing Company, Inc, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Receive between 22 and 29 days of Cutivate lotion treatment
  Fluticasone propionate 0.05% lotion: Daily applications
Period: Overall Study
Arm/Group | Experimental
Started | 56
Completed | 52
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Baseline HPA Axis Supression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.2 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 19
  More than one race | 7
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Post Treatment Serum Cortisol Values Will be Compared.
Description: The primary safety parameter was the response to the CST at the end of treatment/final visit. Blood samples were collected prior to injection of cosyntropin and post-injection. Post-CST stimulation cortisol level ≤ 18micrograms/dL was considered as evidence of adrenal suppression.
Time Frame: Up to 29 days of treatment
Measure: Number; unit: participants
Arm/Group | Experimental
Number analyzed (Participants) | 56
participants | 1

2. Secondary Outcome: Record Skin Atrophy, Pigmentation Change, Hematological and Chemistry Assessments, and Changes in Atopic Dermatitis Severity
Description: The frequency distributions of the presence/absence of adverse events associated with signs of atrophy and pigmentation changes were summarized with frequency counts. Hematology and Chemistry Assessments were summarized in shift tables. Signs and symptoms of AD were summarized at each visit.
Time Frame: Over 5-6 visits following the baseline visit through the end of treatment between Day 22-29
Measure: Number; unit: participants
Arm/Group | Experimental
Number analyzed (Participants) | 56
participants
  skin atrophy | 1
  pigmentation change | 9

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | Experimental
Serious Adverse Events (participants affected / at risk) | 1/56
Other Adverse Events (participants affected / at risk) | 25/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=56)
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=56)
Gastroenteritis (Infections and infestations) | 2 (2)
Herpes simplex (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Folliculitis (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Irritability (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (3)
Ichthyosis (Congenital, familial and genetic disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other